CLINICAL TRIAL: NCT02039765
Title: A Prospective, Single-Center, Open-Label, Study of the Plasma Pharmacokinetics and Safety Following Topical Administration of Brimonidine Tartrate Ophthalmic Solution 0.025% Used Four Times Daily in Healthy, Adult Subjects.
Brief Title: Pharmacokinetics and Safety of Topical Administration of Brimonidine Tartrate Ophthalmic Solution 0.025%.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Collaborators: ORA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 863/13-100-0007
Record Dates: First submitted 2014-01-16; First posted 2014-01-20 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Hyperemia
Keywords: Ocular Redness
MeSH Terms: conditions — Hyperemia | interventions — Brimonidine Tartrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Brimonidine tartrate (Experimental): One drop of brimonidine tartrate ophthalmic solution 0.025% in each eye once at Visit 2 (Day 1) then four times daily (QID) approximately 4 hours apart at Visit 3 (Day 2) through day 6, and then once at Visit 4 (Day 7).
  Interventions: Drug: Brimonidine tartrate

INTERVENTIONS:
Drug: Brimonidine tartrate

SUMMARY:
To characterize the plasma pharmacokinetics and safety profile of brimonidine following a single dose and 4 times per day (QID) dosing of brimonidine tartrate ophthalmic solution 0.025% for 7 days in healthy, adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* have ocular health within normal limits.
* have blood (hematology, blood chemistry) and urine analysis within normal limits.
* have a body weight within 15% of ideal weight

Exclusion Criteria:

* have known contraindications or sensitivity to the use of any of the investigational drug(s) or their components, or any other medications required by the protocol;
* have any active systemic or ocular disorder other than refractive disorder.
* have presence of any abnormality of the lids, ocular surface, or lacrimal duct system that in the Investigator's opinion could affect ophthalmic drop absorption.
* have a history of chronic alcohol consumption.
* consume alcohol and/or caffeine or xanthine containing products within 48 hours prior to dosing at Visit 1 or anticipated use during the study.
* have a history of tobacco, nicotine, or nicotine containing product use within the last year prior to Visit 2;
* have significant weight change (over 10 pounds) within the 60 days prior to Visit 2;
* have blood donation or equivalent blood loss of 450 ml or more, within 60 days prior to Visit 2;
* have an abnormal blood pressure (defined as ≤ 90 or ≥ 160 (systolic) measured in mmHg or ≤ 60 or ≥ 100 (diastolic) measured in mmHg);
* have intraocular pressure (IOP) that is less than 5 mmHg or greater than 22 mmHg or have a normal IOP with a diagnosis of glaucoma.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Plasma Levels | Day 1 (Visit 2)
  Blood samples will be collected for the determination of brimonidine in plasma at the specified time points on Day 1.
Plasma Levels | Day 2 (Visit 3)
  Blood samples will be collected for the determination of brimonidine in plasma at the specified time points on Day 2.
Plasma Levels | Day 7 (Visit 4)
  Blood samples will be collected for the determination of brimonidine in plasma at the specified time points on Day 7.
Plasma Levels | Day 8 (Visit 5)
  Blood samples will be collected for the determination of brimonidine in plasma at the specified time points on Day 8.

SECONDARY OUTCOMES:
Visual Acuity | Baseline (Visit 1)
  Visual acuity testing should be done with best correction at 10ft
Slit Lamp Biomicroscopy | Baseline (Visit 1)
  Lid and lid margin erythema and swelling, conjunctival erythema/hyperemia and chemosis will be graded on a scale of 0 - 4. with 0=normal and 4=marked. Half grade measurements will be accepted for erythema/hyperemia.
Intraocular Pressure | Day 8 (Visit 5)
  Intraocular Pressure measured at baseline Day 8 (Visit 5)
Hematology and Blood Chemistry Analysis | Baseline (Visit 1)
  Blood samples will be collected for hematology and blood chemistry parameters at Baseline (Visit 1)
Urinalysis | Baseline (Visit 1)
  Urine sample will be collected for urinalysis at Baseline (Visit 1)
Visual Acuity | Day 1 (Visit 2)
  Visual acuity testing should be done with best correction at 10ft
Visual Acuity | Day 7 (Visit 4)
  Visual acuity testing should be done with best correction at 10ft
Visual Acuity | Day 8 (Visit 5)
  Visual acuity testing should be done with best correction at 10ft
Slit Lamp Biomicroscopy | Day 1 (Visit 2)
  Lid and lid margin erythema and swelling, conjunctival erythema/hyperemia and chemosis will be graded on a scale of 0 - 4. with 0=normal and 4=marked. Half grade measurements will be accepted for erythema/hyperemia.
Slit Lamp Biomicroscopy | Day 7 (Visit 4)
  Lid and lid margin erythema and swelling, conjunctival erythema/hyperemia and chemosis will be graded on a scale of 0 - 4. with 0=normal and 4=marked. Half grade measurements will be accepted for erythema/hyperemia.
Slit Lamp Biomicroscopy | Day 8 (Visit 5)
  Lid and lid margin erythema and swelling, conjunctival erythema/hyperemia and chemosis will be graded on a scale of 0 - 4. with 0=normal and 4=marked. Half grade measurements will be accepted for erythema/hyperemia.
Intraocular Pressure | Baseline (Visit 1)
  Intraocular Pressure measured at baseline (Visit 1)
Hematology and Blood Chemistry Analysis | Day 8 (Visit 5)
  Blood samples will be collected for hematology and blood chemistry parameters at Day 8 (Visit 5)
Urinalysis | Day 8 (Visit 5)
  Urine sample will be collected for urinalysis at Day 8 (Visit 5)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Ciolino, MD, Study Director — ORA, Inc.
Locations (1):
- Bausch & Lomb, Incorporated, Rochester, New York, United States